CLINICAL TRIAL: NCT05850702
Title: Attenuation of the Hemodynamic Response to Double-lumen Endotracheal Intubation With Nebulized Lidocaine: a Randomized, Double-blind, Controlled Trial
Brief Title: Attenuation of the Hemodynamic Response to Double-lumen Endotracheal Intubation With Nebulized Lidocaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, zhuhao, attending physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIT-2022-0250
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lung Neoplasms
Keywords: Double-lumen Endotracheal Intubation
MeSH Terms: conditions — Lung Neoplasms | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine (Experimental): Intervention group
  Interventions: Drug: Lidocaine
- saline (Placebo Comparator): control group
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — inhale 5ml of 2% lidocaine by nebulization
  Arms: lidocaine
Drug: Saline — inhale 5ml of saline by nebulization
  Arms: saline

SUMMARY:
The goal of this clinical trial is to test the effect of nebulized lidocaine on the hemodynamic response in the participant undergoing double-lumen endotracheal intubation.

The main question it aims to answer is to evaluate the changes in mean arterial pressure after intubation.

Participants will inhale 5ml of 2% lidocaine by nebulization15min before intubation.

Researchers will compare saline group to see if saline effects

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 years, American Society of Anesthesiologists class I-II
2. participants undergoing double-lumen endotracheal intubation under general anesthesia
3. signed informed consent and volunteered to participate in the experiment

Exclusion Criteria:

1. Poor control of hypertension
2. preoperative arrhythmia
3. severe coronary artery or heart valve disease
4. sequelae of cerebrovascular accident
5. severe lung, liver, kidney and immune system diseases
6. Suspected difficult airway
7. confirmed or suspected allergy to this trial drug
8. As judged by the investigator to be ineligible for the study, such as communication impairment (language or intelligence)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
mean arterial pressure after intubation | Immediately after intubation

IPD SHARING:
Plan to Share IPD: No